CLINICAL TRIAL: NCT04742218
Title: A Randomized, Open Label, Two-sequence, Two-period Crossover Study to Assess the Food Effect on the Pharmacokinetics of Single-Dose Administration of the To-Be-Marketed Formulation of K-877 in Healthy Adult Volunteers
Brief Title: Study to Assess the Food Effect of K-877 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: K-877-110
Record Dates: First submitted 2021-01-29; First posted 2021-02-08 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Healthy
MeSH Terms: interventions — K-877 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasted-Fed (Experimental): Single dose of K-877 administered in a fasted condition on Day 1 (Treatment Period 1) and postprandially on Day 4 (Treatment Period 2)
  Interventions: Drug: K-877
- Fed-Fasted (Experimental): Single dose of K-877 administered postprandially on Day 1 (Treatment Period 1) and in a fasted condition on Day 4 (Treatment Period 2)
  Interventions: Drug: K-877

INTERVENTIONS:
Drug: K-877 — K-877 Tablet

SUMMARY:
Study is to assess the effects of food on the Pharmacokinetics(PK) of single-dose administration of K-877 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study-specific evaluation is performed;
* Subject is a healthy adult male or female volunteer between the ages of 18 and 45 years, inclusive, at screening;
* Subject has a BMI of 18 to 30 kg/m2, inclusive, at screening
* Subject meets all inclusion criteria outlined in the clinical study protocol

Exclusion Criteria:

* Subject is a woman who is pregnant or breastfeeding;
* Subject has clinically significant abnormalities in the screening or check-in assessments;
* Subject has received an investigational drug within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug
* Subject does not meet any other exclusion criteria outlined in clinical study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-04-11 (Actual)

PRIMARY OUTCOMES:
Cmax of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Observed maximum plasma concentration (Cmax)
AUC0-t of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Area under the plasma concentration versus time curve from time 0 to the time of the last quantifiable concentration (AUC0-t)
AUC0-inf of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Area under the plasma concentration versus time curve from time 0 extrapolated to infinity (AUC0-inf)

SECONDARY OUTCOMES:
Tmax of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Time to reach the observed maximum (peak) plasma concentration (Tmax)
MRT0-t of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Mean residence time from time 0 to the time of the last quantifiable concentration (MRT0-t)
MRT0-inf of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Mean residence time from time 0 extrapolated to infinity (MRT0-inf)
t1/2 of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Terminal elimination half-life (t1/2)
Kel of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Terminal elimination rate constant (Kel)
CL/F of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Apparent oral clearance (CL/F)
Vd/F of K-877 | pre-dose (within 1 hour before dosing and at pre-meal in case of fed condition) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours after dosing on Days 1 and 4
  Apparent volume of distribution (Vd/F)

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline to Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Shona Pendse, MD, MMSc, Study Chair — Kowa Research Institute, Inc.
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No